CLINICAL TRIAL: NCT06925425
Title: Effect of Task Specific Electrical Stimulation on Upper Limb Gross Motor Skills in Children With Spastic Quadriplegia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Aalaa Farag Soliman, aalaa ahmed farrag, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-420
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy (CP); Spastic Cerebral Palsy; Quadriplegic Cerebral Palsy; Upper Limb Function; Gross Motor Delay
Keywords: TASES; Cerebral palsy; Gross motor skills; Upper limb; Task specific electrical stimulation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Intervention study model Parallel assignment. The study will include thirty children with spastic quadriplegic CP of both sex. Their age will range from two to six years meeting the inclusion criteria will be randomly assigned to two experimental groups : First experimental group: children in this group will receive a designed physical therapy program, attending three sessions per week for three consecutive months. The duration of the session was one hour of the designed physical therapy program. Second experimental group: children in this group will receive the designed program plus the task specific electrical stimulation (TASES) for 20 minutes during the weight bearing exercises as push up , prone on hands on wedge and quadruped with weight shifting.
Masking Description: Intervention study model Parallel assignment. The study will include thirty children with spastic quadriplegic CP of both sex. Their age will range from two to six years meeting the inclusion criteria will be randomly assigned to two experimental groups : First experimental group: children in this group will receive a designed physical therapy program, attending three sessions per week for three consecutive months. The duration of the session was one hour of the designed physical therapy program. Second experimental group: children in this group will receive the designed program plus the task specific electrical stimulation (TASES) for 20 minutes during the weight bearing exercises as push up , prone on hands on wedge and quadruped with weight shifting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) (Experimental)
  Interventions: Other: Designed Physical therapy program
- Group (B) (Experimental)
  Interventions: Other: Task specific electrical stimulation ( TASES ); Other: Designed Physical therapy program

INTERVENTIONS:
Other: Task specific electrical stimulation ( TASES ) — Each child in group B receive the designed program plus the task specific electrical stimulation (TASES) for 20 minutes during the weight bearing exercises as push up , prone on hands on wedge and quadruped with weight shifting.
  The electrical stimulation is applied with the following parameters. Pulse frequency 25-50 HZ, pulse duration 300 micro second, intensity to display a visible muscle contraction, for 20 minutes.
  First channel, one electrode will be placed at the middle of triceps muscle, the second electrode will be placed more distal towards the elbow joint itself (about 3 cm above the olecranon process).
  Second channel, one electrode will be placed over finger and wrist extensors motor point to allow activation of fingers and wrist extensors. The other electrode will be placed over the tendonous portion of the forearm between motor points of extensor carpi radialis and extensor carpi ulnaris muscles.
  Arms: Group (B)
Other: Designed Physical therapy program — The program used a combination of open-and closed-chain exercises. Exercises for facilitating transitions as supine to sit with hand weight bearing , side lying to side sit , side sitting to quadruped, weight bearing exercises as prone on hands on wedge , quadruped with weight shifting and push up exercise for one hour.

SUMMARY:
Cerebral palsy is a non-progressive lesion of the brain occurring before 2 years of age resulting in disorders of posture and movement.( Ostensjo S, 2004)( Keles MN, 2018). Although non- progressive, motor impairments develop as the child grows leading to activity and participation restriction.

For children with CP, body function and structure impairments include changes in muscle tone and strength that affect the ability to control movement, specifically in regard to postural responses, selective control, regulation of activity, ability to learn unique movements, and inappropriate sequencing.(Ross SA,2007)( Ostensjo S, 2004) .

Lack of proper loading and maladaptive muscle pulls over time causes the skeletal system to adapt to positions of malalignment, malformation, and overall bone weakness (Beckung E, 2007) (Elbasan B, 2018).

These changes lead to delays in the natural progression of gross motor skills. As the child falls behind in motor function, they also fall behind in cognitive stimulation and development.( Akaya KU, 2018) . Understanding the anatomical and physiological implications that CP has on the developing child is necessary for physical therapists to treat this population, especially when utilizing electrical stimulation.

Spastic quadriplegia Is a type of cerebral palsy that affects all four limbs and typically involves significant motor impairment. It results from brain damage that occurs before, during, or shortly after birth, affecting the areas of the brain responsible for movement and coordination.

Electrical stimulation is a mode of physical therapy that can be utilized in the treatment of various nerve and muscle injuries, in addition to patients with acute and chronic pain. It involves an electrical pulse applied to a muscle or nerve that activates excitable tissue utilizing internal or external electrodes to build muscle strength, reduce pain, as well as create or support limb movement (Kerr C, 2007).

Task-specific electrical stimulation (TASES) is a therapeutic technique used primarily in rehabilitation settings to enhance motor function. The primary aim of TASES is to facilitate movement and improve motor learning by applying electrical stimulation to specific muscles during targeted tasks.

DETAILED DESCRIPTION:
Cerebral palsy is a group of non-progressive motor disorders; it commonly appears in early childhood and affects muscle tone, posture, and movement. (Salazar AP, 2019) The most common cause of physical disability in developed countries and one of the most common causes of acquired physical disability in children is cerebral palsy (Surveillance of cerebral palsy in Europe, 2000). between 1.5 and 4 per 1000 live births, on average (Smithers-Sheedy H, 2016).An estimated 17 million people live with cerebral palsy worldwide, and at least 80 percent of them will survive into their sixth decade ( Blair E, 2019).

This definition acknowledged that there are numerous etiologies for cerebral palsy and that, although the movement and posture disorders are permanent, the motor impairments are frequently progressive.

Classification in CP uses different descriptors and may assess different aspects of the clinical manifestation such as topography of affected limbs, severity of movement impairment, or upper limb manual ability. For instance, regarding topographical classification, unilateral involve- ment of an arm and leg is termed hemiplegia, predomi- nant lower limb involvement is termed diplegia, and involvement of all limbs is termed quadriplegia (Shevell MI, 2010) (Stanley FJ,2000).

Tone abnormalities result from the area of the central nervous system that is damaged. Damage at the vestibulospinal and rubrospinal pathways of the spinal cord and associated central cortex of the brain, accounting for 80% of cases, results in spasticity, at the basal ganglia results in dyskinesia, at the cerebellum results in ataxia, or a mix of any of these.( Goodman CC, 2015) Damage to the cortex, can result in the topography presentations of monoplegia, hemiplegia, diplegia, or quadriplegia, and at the basal ganglia athetoid. ( Ko, N.2022)

Spastic quadriplegia is a type of cerebral palsy characterized by increased muscle tone and stiffness affecting all four limbs, often resulting in significant motor impairment. (Smith J, 2023)

Key Features:

1. Motor Impairment: Individuals may have severe limitations in movement and muscle control, impacting their ability to walk or use their hands.
2. Muscle Tone: Muscle tone can vary, leading to stiffness (spasticity) or weakness. This can affect posture and mobility.
3. Associated Conditions: Many individuals with quadriplegic cerebral palsy may also experience other challenges, such as intellectual disabilities, seizures, or sensory impairments. (Rosenbaum P, 2007)

Upper limb problems in individuals with spastic quadriplegia can vary widely, but some common issues include:

1. Muscle Tone and Spasticity: Muscles in the arms may be excessively tight, leading to difficulty in movement. This spasticity can cause awkward positioning of the hands and arms.
2. Limited Range of Motion: Joint stiffness, particularly in the shoulders, elbows, and wrists, can restrict the range of motion. This can make it challenging to perform everyday tasks.
3. Weakness: While spasticity affects muscle tone, many individuals also experience muscle weakness, which can impact the ability to grasp, lift, or manipulate objects.
4. Postural Issues: Poor posture can further complicate upper limb function. Malalignment of the shoulders or spine can affect how well the arms can be used.
5. Fine Motor Skills: Difficulties with fine motor skills can impede activities such as writing, using utensils, or buttoning clothing.
6. Sensory Issues: Some individuals may also have sensory processing issues, making it hard to feel objects or differentiate between textures.
7. Contractures: Over time, muscle tightness can lead to contractures, where joints become permanently bent, further limiting function.
8. Pain and Discomfort: Spasticity and muscle imbalances can lead to discomfort or pain in the upper limbs.

(Smith J, 2023) Upper limb gross motor skills involve the use of larger muscle groups to perform movements that require coordination and balance, such as reaching, lifting, and throwing. In individuals with spastic CP, these skills can be impaired in several ways.

Key Impacts on Upper Limb Gross Motor Skills :

1. Spasticity:

   Muscle Tone: Increased muscle tone leads to stiffness, making it difficult to initiate and control movements. This can result in awkward postures, such as flexed elbows or wrists.

   Movement Patterns: Movements may become jerky or uncoordinated, making activities like reaching or throwing difficult.
2. Limited Range of Motion:

   Joint Stiffness: Tightness in muscles and tendons can restrict the range of motion in the shoulders, elbows, and wrists, affecting the ability to perform full movements. Contractures: Over time, muscle tightness can lead to permanent shortening (contractures), further limiting function.
3. Poor Coordination and Control: Proprioception: Difficulty in sensing body position can impact the ability to coordinate arm and hand movements effectively.
4. Balance Issues: Poor balance can affect the stability required to use the arms for gross motor tasks, such as throwing a ball or climbing.
5. Postural Control:

Core Stability: Good upper limb function often depends on a stable trunk. Weak core muscles can make it harder to control arm movements during activities.

Alignment: Abnormal postures can affect how the arms are used, leading to compensatory strategies that are less effective. (Smith J, 2023)

Upper limb and gross motor skills and postural mechanisms:

1. Establish head control (stability and movement) for hand/eye coordination.
2. Establish postural stability and weight shift of head, shoulder girdle, trunk and pelvis in many gross motor activities in prone, supine, sitting, standing and stepping, which are also necessary for hand function. This allows arm and hand function in postures other than in lying.
3. Develop rising reactions. Hands and arms are used to help in the change of various postures or the assumption of posture in gross motor development. A child also needs to assume a position in which he will carry out his chosen task in various environments.
4. Develop saving reactions in the arms. The up- per limbs are thrown into various patterns in- volving active contractions of the muscles in synergies (patterns) to save and prop the child as he falls off balance.
5. Some of the arm synergies trained for gross motor function are also used in voluntary reach. (Levitt S. 2010)

Task-Specific Electrical Stimulation (TASES) Definition TASES involves applying electrical stimulation to muscles during the performance of specific tasks or movements. The goal is to improve motor function, enhance muscle activation, and facilitate motor learning.

Mechanism

* Electrical Stimulation: Electrodes are placed on the skin over the targeted muscles. Electrical impulses stimulate muscle contractions.
* Task-Specific Context: The stimulation is synchronized with task performance, meaning the muscles are activated when the patient is attempting to perform a specific movement, like reaching or grasping. (Cramer SC 2012)

Benefits:

* Motor Learning: By pairing electrical stimulation with functional tasks, TASES helps reinforce neural pathways associated with those movements.
* Strengthening: It can improve muscle strength and endurance in targeted areas.
* Improved Coordination: Helps enhance the coordination and timing of muscle contractions.
* Functional Independence: Aims to increase the ability of individuals to perform daily activities more independently. (Dario C,2016)

Key Components of TSES:

1. Targeted Muscle Activation: TSES involves applying electrical stimulation to muscles that are involved in specific tasks, such as grasping, walking, or reaching. This helps to activate muscles that may not be functioning optimally due to injury.
2. Task-Specific Training: The stimulation is synchronized with the performance of specific tasks. This can help reinforce neural pathways associated with those movements, promoting better motor control and learning.
3. Neuroplasticity: By pairing electrical stimulation with motor tasks, TSES can enhance neuroplasticity, the brain's ability to reorganize itself and form new neural connections. This is crucial for recovery in post-stroke rehabilitation.
4. Functional Outcomes: Research has shown that TSES can improve functional outcomes, such as increased strength, improved coordination, and greater independence in daily activities.
5. Customization: TSES protocols can be tailored to individual patients, considering factors like the specific muscles involved, the type of injury, and the rehabilitation goals. (Smith J, 2023)

Children's gross motor function has a direct impact on quality of life metrics like participation and activity (Palisano RJ, 2009). Children with cerebral palsy (CP) frequently experience difficulties with their gross motor skills (Rosenbaum PL, 2002).

Maximizing functional abilities is a key objective of treatment for these children. Because of limited research area to evaluate the relation between gross motor skills with the upper limb muscles strength therefore, the aim of the current study is to investigate this relation.

It is commonly recognized that the two main issues seen in children with CP are a delayed development of gross motor function and a decline in postural control. As a result, children with spastic cerebral palsy are unable to carry out a number of daily tasks, such as standing, sitting, and walking. For many functional activities, the ability to sit is crucial because it makes transfers easier and permits independent upper limb manipulation of objects. (Beckung E, 2007) (Akaya KU, 2018).

ELIGIBILITY:
Inclusion Criteria:

1. Their age will be ranged from 2 to 6 years. Their grade of spasticity will be from 1+ to 2 according to Modified Ashworth scale (Baunsgaard etal., 2016). (APPENDIX II).
2. They will be on Level III and IV according to Gross Motor Functional Classification System (GMFCS) (Palisano et al., 2008).(APPENDIX III).
3. Parents/legals representatives consenting to their child's participation 5 - Diagnosed with Spastic Quadriplegic cerebral palsy

Exclusion Criteria:

1. Previous neurological or orthopedic surgery in the upperextremities.
2. Fixed deformity in the joints of upper limb. 3- Severe hearing and visual defect.

4-Irregular attendance at assessments or therapy sessions

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Improved upper limb gross motor skills | after 3 months of treatment
  The Quality of Upper Extremity Skills Test (QUEST) is used by assessment of the weight bearing domain .

SECONDARY OUTCOMES:
Improvement in joints range of motion | after 3 months of treatment
  Electronic Digital Goniometer will be used in this study to measure ROM of wrist and elbow extension .

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bedair Ibrahim, professor of physical therapy, Principal Investigator — kafr-elsheikh university
Locations (1):
- Aalaa Ahmed Farrag, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided